CLINICAL TRIAL: NCT03181542
Title: A Randomized Controlled Study of Efficacy of Infra Red Vein Illumination Versus Standard Technique
Brief Title: Infra Red Vein Visualization: Efficacy vs. Standard Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Priti G. Dalal, Professor of Anesthesiology & Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00006768
Record Dates: First submitted 2017-06-01; First posted 2017-06-08 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: Difficult Intravenous Access

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Infrared vein illumination (Experimental): Infrared illumination of veins, using the FDA approved AccuVein device, will be used to assist in vein location when inserting an intravenous access line
  Interventions: Device: Infrared illumination
- Standard Technique (No Intervention): Standard vein location techniques will be used when inserting an intravenous access line

INTERVENTIONS:
Device: Infrared illumination — Infrared illumination of veins using the FDA approved AccuVein (AccuVein, Inc., Huntington, NY) device.
  Arms: Infrared vein illumination

SUMMARY:
The objective of the study is to assess the efficacy of the vein visualization device AccuVein (AccuVein, Inc., Huntington, NY) in comparison to a standard technique for establishing intravenous (iv) access in the infant and toddler population (<2years)

DETAILED DESCRIPTION:
The objective of this project is to compare the iv success rate using the FDA approved Accuvein device for vein illumination versus not using the device, for infants/toddlers undergoing surgery at Penn State Children's Hospital with an ASA physical status 1, 2, or 3. After obtaining informed consent, the infant will be randomized to the vein illuminatin or standard group based on a computer generated number.

ELIGIBILITY:
Inclusion Criteria:

1. Children(<2year) undergoing anesthesia procedures at Penn State Health, Hershey Medical Center and Penn State Children's Hospital
2. ASA physical status 1,2 or 3

Exclusion Criteria:

1. Emergency procedures requiring anesthesia
2. ASA physical status 4
3. Patients with pre existing iv access

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priti G Dalal, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaddoum RN, Anghelescu DL, Parish ME, Wright BB, Trujillo L, Wu J, Wu Y, Burgoyne LL. A randomized controlled trial comparing the AccuVein AV300 device to standard insertion technique for intravenous cannulation of anesthetized children. Paediatr Anaesth. 2012 Sep;22(9):884-9. doi: 10.1111/j.1460-9592.2012.03896.x. Epub 2012 Jun 14. PMID 22694242
- [Background] Rothbart A, Yu P, Muller-Lobeck L, Spies CD, Wernecke KD, Nachtigall I. Peripheral intravenous cannulation with support of infrared laser vein viewing system in a pre-operation setting in pediatric patients. BMC Res Notes. 2015 Sep 21;8:463. doi: 10.1186/s13104-015-1431-2. PMID 26391665
- [Background] de Graaff JC, Cuper NJ, Mungra RA, Vlaardingerbroek K, Numan SC, Kalkman CJ. Near-infrared light to aid peripheral intravenous cannulation in children: a cluster randomised clinical trial of three devices. Anaesthesia. 2013 Aug;68(8):835-45. doi: 10.1111/anae.12294. Epub 2013 Jun 14. PMID 23763614
- [Background] Nafiu OO, Burke C, Cowan A, Tutuo N, Maclean S, Tremper KK. Comparing peripheral venous access between obese and normal weight children. Paediatr Anaesth. 2010 Feb;20(2):172-6. doi: 10.1111/j.1460-9592.2009.03198.x. Epub 2009 Nov 17. PMID 19922428
- [Background] Jacobson AF, Winslow EH. Variables influencing intravenous catheter insertion difficulty and failure: an analysis of 339 intravenous catheter insertions. Heart Lung. 2005 Sep-Oct;34(5):345-59. doi: 10.1016/j.hrtlng.2005.04.002. PMID 16157191
- [Background] Yen K, Riegert A, Gorelick MH. Derivation of the DIVA score: a clinical prediction rule for the identification of children with difficult intravenous access. Pediatr Emerg Care. 2008 Mar;24(3):143-7. doi: 10.1097/PEC.0b013e3181666f32. PMID 18347490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects will be identified from the electronic operating room scheduling system (surginet) by reviewing the operative list schedule the day before or on the day of their scheduled surgical or diagnostic procedure.
Period: Overall Study
Arm/Group | Infrared Vein Illumination | Standard Technique
Started | 80 | 80
Completed | 79 | 80
Not Completed | 1 | 0
Not completed — Subject withdrawn because research physician could not make it in time to place IV | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infrared Vein Illumination | Standard Technique | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.11 (6.19) | 12.42 (6.44) | 12.76 (6.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 38 | 74
  Male | 43 | 42 | 85
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 60 | 56 | 116
  African American | 5 | 8 | 13
  Hispanic/Latino | 8 | 10 | 18
  Asian | 2 | 2 | 4
  Mixed Race | 3 | 2 | 5
  Other | 1 | 1 | 2
  Unknown | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 79 | 80 | 159
Skin Color [Count of Participants; unit: Participants] — Population: Skin color data was not collected from 1 standard subject
  Participants
    number analyzed (Participants) | 79 | 79 | 158
    Light | 60 | 57 | 117
    Medium | 15 | 18 | 33
    Dark | 4 | 4 | 8
Anticipated IV access difficulty [Number; unit: participants] — Anticipated IV access difficulty is scored on a subjective Likert Scale where 0 is no anticipated difficulty and 5 is extreme anticipated difficulty Population: Data was not collected for the anticipated IV access difficulty for 1 standard subject
  participants
    0: number analyzed (Participants) | 79 | 79 | 158
    0 | 0 | 5 | 5
    1: number analyzed (Participants) | 79 | 79 | 158
    1 | 14 | 9 | 23
    2: number analyzed (Participants) | 79 | 79 | 158
    2 | 22 | 19 | 41
    3: number analyzed (Participants) | 79 | 79 | 158
    3 | 23 | 26 | 49
    4: number analyzed (Participants) | 79 | 79 | 158
    4 | 11 | 11 | 22
    5: number analyzed (Participants) | 79 | 79 | 158
    5 | 9 | 9 | 18
Prematurity [Count of Participants; unit: Participants] — Prematurity is defined as live birth prior to 37 weeks gestation Population: Prematurity data was not entered for 1 Infrared vein illumination subject
  Participants
    number analyzed (Participants) | 78 | 80 | 158
    yes | 13 | 12 | 25
    no | 65 | 68 | 133
ASA physical Status [Count of Participants; unit: Participants] — ASA1=healthy patients ASA2=mild to moderate systemic disease caused by the surgical condition or by other pathological processes, and are medically well controlled ASA3=severe disease process which limits activity but is not incapacitating ASA4=severe disease process that is a constant threat to life ASA5=moribund patient not expected to survive 24 hours with or without an operation ASA6=Declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    1 | 19 | 21 | 40
    2 | 47 | 43 | 90
    3 | 13 | 16 | 29
    4 | 0 | 0 | 0
    5 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] | 9.45 (2.32) | 9.13 (2.23) | 9.30 (2.28)
Time without liquids [Mean (Standard Deviation); unit: hours] | 6.93 (3.82) | 6.37 (3.72) | 6.66 (3.77)

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Success for insertion of intravenous access line will be determined by flushability with 5 ml of sterile normal saline
Time Frame: When patient is in operating room and insertion of intravenous access line has been confirmed to be successful, an average of 30 minutes
Measure: Number; unit: percentage of participants
Arm/Group | Infrared Vein Illumination | Standard Technique
Number analyzed (Participants) | 79 | 80
percentage of participants | 84.81 | 90
Statistical Analysis 1: Comparison: Infrared Vein Illumination vs Standard Technique; Test type: Superiority; p = 0.34, Fisher Exact

2. Secondary Outcome: The Number of Attempts
Description: The number of attempts it takes for successful insertion of the intravenous access line
Time Frame: When patient is in operating room and insertion of intravenous access line is performed
Measure: Mean (Standard Deviation); unit: number of attempts
Arm/Group | Infrared Vein Illumination | Standard Technique
Number analyzed (Participants) | 79 | 80
number of attempts | 1.93 (1.46) | 2.15 (3.11)
Statistical Analysis 1: Comparison: Infrared Vein Illumination vs Standard Technique; Test type: Superiority; p = 0.40, Jonckheere-Terpstra Test

3. Secondary Outcome: Time to Successful Insertion
Description: The time to successful insertion of the intravenous access line will be measured from the first time that the canula touches the skin to until successful iv access is established
Time Frame: When patient is in operating room and insertion of intravenous access line is performed
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Infrared Vein Illumination | Standard Technique
Number analyzed (Participants) | 79 | 80
seconds | 149.39 (354.04) | 136.92 (179.79)
Statistical Analysis 1: Comparison: Infrared Vein Illumination vs Standard Technique; Test type: Superiority; p = 0.90, Jonckheere-Terpstra Test

ADVERSE EVENTS:
Time Frame: During the procedure up to their discharge from Post-anesthesia care unit or recovery unit up to 1 hour after the procedure, an average of 3 hours total
Arm/Group | Infrared Vein Illumination | Standard Technique
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/80
Other Adverse Events (participants affected / at risk) | 0/79 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT03181542/Prot_SAP_000.pdf